CLINICAL TRIAL: NCT07261033
Title: Exploring the Effectiveness of Equine Assisted Psychotherapy on the Emotional Regulation and Mental Wellbeing of Service Users in an Inpatient Setting Who Have Received a Diagnosis of Emotionally Unstable Personality Disorder
Brief Title: Exploring Equine-Assisted Psychotherapy as an Intervention for Those Who Have Received a Diagnosis of Emotionally Unstable Personality Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cygnet Healthcare (Other)
Collaborators: Track Clinic, Frome (Unknown)
Responsible Party: Principal Investigator, Lewis Byrne, Assistant Psychologist, Cygnet Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 364995
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Emotionally Unstable Personality Disorder, Borderline Type
Keywords: Personality Disorder; Equine Assisted Psychotherapy
MeSH Terms: conditions — Personality Disorders | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Equine-Assisted Psychotherapy (Experimental): All participants will attend 6 half-day sessions of Equine-Assisted Psychotherapy. This is a type of psychotherapy in which the professional(s) and the client(s) are joined by an equine. This will be conducted at a specialist clinic by a member of their facilitator team. There will also be hospital staff on-hand to provide support if needed, but they will not be involved in the therapy directly.
  The therapy will involve a group session (1 hour and 15 minutes long), and individual sessions (30 minutes per participant).
  Interventions: Behavioral: Equine-Assisted Psychotherapy

INTERVENTIONS:
Behavioral: Equine-Assisted Psychotherapy — All participants will attend 6 half-day sessions of Equine-Assisted Psychotherapy. This is psychotherapy between the professional(s) and the client(s) which takes place in the presence of an equine (e.g. horse, alpaca). This will be conducted at a specialist clinic by a member of their facilitator team. There will also be hospital staff on-hand to provide support if needed, but hospital staff will not be involved in the therapy directly. The therapy will involve a group session (1 hour and 15 minutes long), and individual sessions (30 minutes per participant).

SUMMARY:
The purpose of this research is for the multi-disciplinary team at an inpatient psychiatric hospital to investigate more innovative ways to engage service users in order to promote wellbeing and emotional regulation. In particular, there is a focus on engaging patients who do not routinely engage with the Psychology Team. As such, we are aiming to explore the effectiveness of Equine Assisted Psychotherapy (EAP) with the service users on a specialist Personality Disorder ward.

EAP is the deliberate inclusion of an equine (e.g. horse, alpaca) amongst a therapy team to improve patient outcomes. This therapy team includes a mental health professional and certified equine specialist, along with equine(s) and client(s). EAP can offer specific psychotherapeutic treatment goals such as addressing trauma and emotion dysregulation. The presence of an equine removes the need for verbal communication, which allows for non-verbal approaches that support self-development; identifying and discussing the feelings, emotions and behaviours generated through interaction with the horse. The presence of equine also provides a unique opportunity for traumatised individuals to build trust with other sentient beings that value connection, safety, and trust.

These specific psychotherapeutic treatment goals are especially relevant for those with a diagnosis of Emotionally Unstable Personality Disorder (EUPD). Service users with EUPD present with complex mental health difficulties, often with problems with emotional regulation, attachment, and self-harm.

This research will use a qualitative, single arm design in which all participants (inpatients who have received an Emotionally Unstable personality Disorder diagnosis) engage in a novel psychotherapeutic intervention (6 sessions of Equine-Assisted Psychotherapy). Their experiences of this psychotherapeutic intervention will be explored using semi-structured interviews. Researchers and participants will collaborate in using Thematic Analysis to analyse the content of these interviews.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient on the ward (name of ward not included for confidentiality).
* Has received a diagnosis of Emotionally Unstable Personality Disorder.
* Since participants will be under Section 3 of the Mental Health Act, they must have the required Section 17 therapy leave at the time of recruitment.
* Service users will have been assessed for their capacity to consent by the Multi-Disciplinary Team and deemed to have capacity at the time of recruitment.
* All participants on the ward are female and between 18-65.

Exclusion Criteria:

* If the Multi-Disciplinary Team's assessment is that they do not have capacity to consent.
* Those who do not have the relevant Section 17 leave.
* Patients who have a planned discharge date that is before the intended end date of the research.
* Patients who have previous experience with Equine Assisted Psychotherapy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Perception of Emotional Regulation | From enrolment to 1 week after end of last Equine-Assisted Psychotherapy session. This should be a maximum of 8 weeks in total.
  This will be measured via semi structured interview questions and the thematic analysis of participants' responses. It will focus on whether participants notice a difference in how they are able to regulate their emotions following therapeutic intervention and, if so, what that change is and why participants think that change has happened.
Perception of Connection to Others | From enrolment to 1 week after end of last Equine-Assisted Psychotherapy session. This should be a maximum of 8 weeks in total.
  This will be measured via semi structured interview questions and the thematic analysis of participants' responses. It will focus on whether participants notice a difference in how they are able to connect with others following therapeutic intervention and, if so, what that change is and what they think caused it.
General Experience of Therapeutic Intervention | From first therapy session to one week after the last Equine-Assisted Psychotherapy session. Up to 7 weeks in total.
  This will be measured via semi structured interview questions and the thematic analysis of participants' responses. It will focus on how the participants felt about the therapy e.g. what they liked/disliked about it and which aspects were meaningful to them.
Perception of how Equine-Assisted Psychotherapy compares to other therapies. | From first therapy session to one week after the last Equine-Assisted Psychotherapy session. Up to 7 weeks in total.
  This will be measured via semi structured interview questions and the thematic analysis of participants' responses. It will focus on how the participants felt this therapy compared to other therapies they have experience e.g. In what ways is it better/worse?

SECONDARY OUTCOMES:
Intervention Retention Rate | From start of first Equine-Assisted Psychotherapy session to end of last Equine-Assisted Psychotherapy session. The Equine-Assisted Psychotherapy runs for 6 weeks in total.
  The number of participants that withdraw from the intervention.
Intervention Attendance | From start of first Equine-Assisted Psychotherapy session to end of last Equine-Assisted Psychotherapy session. These run for 6 weeks in total.
  The number of Equine-Assisted Psychotherapy sessions each participant attends.

CONTACTS AND LOCATIONS:
Locations (1):
- Cygnet Hospital Kewstoke, Weston-super-Mare, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No